CLINICAL TRIAL: NCT06633367
Title: Nature Dose Equity for Students
Brief Title: Nature IDEAS Study: An RCT to Increase Time Spent in Nature Among University Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Michigan State University (Other)
Collaborators: Cleveland State University (Other); Clemson University (Other); University of Virginia (Other); University of Maryland (Other); University of Maryland Eastern Shore (Other); Morgan State University (Other); University of New Mexico (Other); North Carolina Agricultural and Technical University (Other); REI Cooperative Action Fund (Unknown); Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Amber Pearson, Associate Professor, Michigan State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: STUDY00010829
Record Dates: First submitted 2024-10-07; First posted 2024-10-09 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Mental Health
Keywords: Mental Health; Nature; Young Adults
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: The investigators will determine nature opportunities at each school using park and sports field mapping, remote sensing, and tree canopy assessment within 30 miles of campuses to identify disparities. As Fall semester starts, the investigators will recruit 160 students/school for an RCT. Students will complete baseline surveys on nature connectedness, nature belongingness, mental health, and demographics. Students will download the NatureDose™ app, which uses 30+ datasets and machine learning models to quantify nature. The app calculates how much nature is near users whenever they are outdoors, and weekly minutes in nature. App data will be collected over a 2-week baseline period, after which students will be randomized to receive 1) standard information about the health benefits of nature or 2) standard health information, a request to increase time in nature, eligibility to receive a prize, and information on peer performance. After 2 weeks, students will repeat baseline surveys.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group receiving standard health information (No Intervention): This group will receive information about health benefits in nature.
- Intervention Group receiving standard health information + incentives to increase time outdoors (Active Comparator): This group will receive information on the health benefits of time outdoors, a request to increase their time outdoors, eligibility to receive a prize, and information on peer performance.
  Interventions: Other: Increasing time in nature

INTERVENTIONS:
Other: Increasing time in nature — This intervention includes requesting an increase in time spent outdoors, eligibility to receive a prize, and information on peer performance.
  Arms: Intervention Group receiving standard health information + incentives to increase time outdoors

SUMMARY:
This project will first examine nature opportunities, belonging and benefits with a multi-state nature-based intervention with a focus on students of color. In light of the syndemic, 'nature deficit disorder' and poor mental health, the investigators anticipate several far-reaching impacts that will (a) test a nationally useful standardized way to quantify exposure; (b) invest in nature resources and accessibility on campuses; and (c) promote the mental health and therapeutic benefits of nature among young adults. These will lead to understanding the nature exposure and mental health interplay and techniques for quantifying and encouraging nature exposure to treat the on-going youth mental health crisis. Including HBCUs and an hispanic-serving institution is expected to result in heightened visibility of underlying disparities, including structural racism and land-based violence and discrimination, that have contributed to current-day nature gaps and dismantled nature relationships for students of color.

DETAILED DESCRIPTION:
America faces a syndemic of youth 'nature deficit disorder' and poor mental health. These conditions can be improved by nature contact, but the outdoors is not equally accessible, particularly for students of color. This study leverages the NatureDose™ app to identify racial/ethnic inequities in nature opportunities, belonging, and benefits and conduct an RCT to improve mental health and address disparities by getting university students outdoors into nature. The investigators will test 3 over-arching questions:

1. Are there differences in nature opportunities and/or belongingness for White versus students of color?
2. Does more time in nature correlate with greater feelings of nature connectedness, belongingness, and better mental health?
3. Is a nature-based intervention that leverages NatureDoseTM a cost-effective way to improve mental health, particularly for students of color?

This project has two stages. 1) We will determine nature opportunities at each institution using park and sports field mapping, remote sensing, and tree canopy assessment within 30 miles of campuses to identify disparities. 2) As Fall semester starts, we will recruit 160 students/site for a randomized controlled trial (N=1,440 total, giving 80% power to detect effects down to Cohen's d=0.2 even with attrition). Students will complete baseline surveys on nature connectedness (NR-6), nature belongingness (validated scale for university students), mental health (distress, worry, positive/negative affect), and demographics. Next, students will download the NatureDose™ app, which uses 30+ datasets and machine learning models to quantify nature. The app calculates how much nature is near users whenever they are outdoors, and weekly minutes in nature. App data will be collected over a 2-week baseline period, after which students will be randomized to receive 1) standard information about the health benefits of nature (50%) (Active Control) or 2) standard health information, a request to increase weekly minutes in nature, eligibility for a prize, and peer performance comparison. After 2 weeks, students will repeat baseline surveys.

ELIGIBILITY:
Inclusion Criteria:

* Undergraduate student
* 18-24 years of age
* Lives within 30 miles of university campus

Exclusion Criteria:

* Not an undergraduate student
* Under 18 or over 24 years of age
* Lives > 30 miles from the university campus

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1545 (Actual)
Dates: Start 2024-09-09 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
Kessler-6 | From enrollment to end of participation phase, 4 weeks.
  Kessler-6 changed to be a two week recall period. Range: 0-24. Higher scores indicate higher distress.
Worry | from enrollment to the final survey (4 week period)
  Single question "I worry all the time" on a likert-type scale. Source: https://pubmed.ncbi.nlm.nih.gov/29214862/. Values range from 1-5, whereby a higher score indicates more frequent worry.
Positive and Negative Affect Scale | from emrollment to the final survey (4 week period)
  This scale is comprised of 20 items, with 10 items measuring positive affect (e.g., excited, inspired) and 10 items measuring negative affect (e.g., upset, afraid). Each item is rated on a five-point Likert Scale, ranging from 1 = Very Slightly or Not at all to 5 = Extremely, to measure the extent to which the affect has been experienced, over a two-week period. Positive affect range: 10-50, whereby higher values indicate higher positive affect. Negative affect range: 10-50, whereby higher values indicate higher negative affect.

SECONDARY OUTCOMES:
NR-6 | From enrollment to the final survey (4 week period)
  Nature relatedness scale, developed by Nisbet and Zelenski. Each question asked on a likert-type scale from 1 to 5. Then these values are averaged (after considering reverse scored items) to create a score (final score range 1-5), whereby higher values indicate higher nature relatedness.
Access to Nature scale | from enrollment to the final survey (4 week period)
  Access to nature scale, developed by Anders et al. Source: https://www.sciencedirect.com/science/article/pii/S0272494422001943#appsec1. There twelve questions employ a Likert-type scale where 1 reflected little-to-no barrier and 5 reflected the greatest barrier to access. All items were reverse scored for a total sum that reflected participants' overall access to nature, whereby higher scores indicate fewer barriers to access (range 12-60).

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - Morgan State University, Baltimore, Maryland
  - University of Maryland, College Park, Maryland
  - University of Maryland Eastern Shore, Salisbury, Maryland
  - Michigan State University, East Lansing, Michigan
  - University of New Mexico, Albequerque, New Mexico
  - North Carolina A&T University, Greensboro, North Carolina
  - Cleveland State University, Cleveland, Ohio
  - Clemson University, Clemson, South Carolina
  - University of Virginia, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: No